CLINICAL TRIAL: NCT05084326
Title: Engagement of Fetal Head as a Predictor of a Successful Vaginal Delivery in Primigravidas Presented in Early Labor
Status: Completed | Type: Observational
Sponsor: mohamed abosena (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Sponsor-Investigator, mohamed abosena, Principal Investigator, Ain Shams University
Organization: Ain Shams University (Other)
Other Study IDs: AinShamsU Hos
Record Dates: First submitted 2021-10-03; First posted 2021-10-19 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Labor Onset and Length Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mohamedabosena
  Interventions: Procedure: Engagement of fetal head as a predictor of a successful vaginal delivery

INTERVENTIONS:
Procedure: Engagement of fetal head as a predictor of a successful vaginal delivery — In addition to the fetal lie, presentation, and position, the level or station of the presenting part in the maternal pelvis is an important factors in the labor process.
  In primigravida, Delayed engagement of fetal head has been theorized that it is more likely in women with a possible cephalo-pelvic disproportion, so far they are associated with higher risk of cervical dystocia, which led to increased rate of caesarean section.

SUMMARY:
In primigravida, Delayed engagement of fetal head has been theorized that it is more likely in women with a possible cephalo-pelvic disproportion, so far they are associated with higher risk of cervical dystocia, which led to increased rate of caesarean section.

DETAILED DESCRIPTION:
This study will involve total 226 of " 113 primigravida patients with engaged head and 113 primigravida patients with unengaged head .

while assessment of fetal head station, status of membrane should be evaluated and noted.

Engagement will be assessed by vaginal examination as described by Müller in 1868 , assumes that when the leading edge of the vertex is felt at the level of the ischial spines, the biparietal diameter will have just passed through the pelvic brim. The leading edge of the vertex at the level of the ischial spines is designated as being at station 0. If the leading edge is 1 cm below the level of the spines, this is referred to as station +1. Usually, a head on the pelvic floor is at station +4 or +5.

Uengaged head is still 2 cm above the level of the spines is at station -2, and so on.

The aim of this study will be to determine if primigravida patients with unengaged head after spontaneous onset of labor are at increased risk of cesarean section.

The patients will be admitted in the labour room. Name, age and detailed history will be noted A thorough general examination and systemic examination will be done to determine the fundal height, the baby's lie, presentation, position, engagement of the presenting part, and frequency and duration of contractions, auscultation of the fetal heart rate for a minimum of 1 minute immediately after a contraction.

A vaginal examination will be offered for more assessment of pelvic status, cervical dilation (in cm) and effacement, position of fetal head and status of membrane will be evaluated and noted.

Assessment of labor progress will be done by digital examination : to document cervical dilation, effacement, and fetal station are usually routinely performed:

* At four hour intervals in the first stage
* Prior to administering analgesia/anesthesia*
* When the parturient feels the urge to push (to determine whether the cervix is fully dilated)
* At one hour intervals in the second stage
* If fetal heart rate abnormalities occur " to evaluate for complications such as cord prolapse "

  * All patients should be counselled and offered Epidural anesthesia during first and second stage of labor.

Observations during the established frst stage:

1. Half-hourly documentation of frequency of contractions
2. Hourly pulse
3. 4-hourly temperature and blood pressure
4. A vaginal examination 4-hourly or if there is concern about progress

If delay is established in first stage of labour of cervical dilatation of less than 2 cm in 4 hours for frst labour , amniotomy should be considered for all women with intact membranes increase the strength and pain of contractions, in normally progressing labour, do not perform amniotomy routinely.

vaginal examination 2 hours later, and diagnose delay if progress is less than 1 cm.

increase the strength and pain of contractions, vaginal examination 2 hours later, and diagnose delay if progress is less than 1 cm.

Decision about management options of oxytocin augmentation according NICE guidelines should considered.

According to RCOG guidelines, we will use a low-dose protocol for all patients, by adding 10 IU oxytocin to 1 litre of 0.9% normal saline.

Electronic fetal monitoring will be performed for a minimum of 20 minutes before starting oxytocin, and will be continued until the baby is delivered, intervention will be according to interpretation of CTG.

According to NICE guidelines, vaginal examination 4 hours after starting oxytocin in established labour:

* If cervical dilatation has increased by less than 2 cm after 4 hours of oxytocin, further obstetric review is required to assess the need for caesarean section.
* If cervical dilatation has increased by 2 cm or more, advise 4-hourly vaginal examinations.

Observations during the second stage:

1. Half-hourly documentation of the frequency of contractions.
2. Hourly blood pressure.
3. Continued 4-hourly temperature.
4. Frequency of passing urine .
5. A vaginal examination hourly in the active second stage.

ELIGIBILITY:
Inclusion Criteria:

* Term pregnancy (37-42) weeks.
* Expected foetal birth weight of 2.5-4.0 kg on USG at term.
* Singleton live pregnancy.
* Cephalic presentation.
* Cervical dilatation of =/< 4cms.
* Reactive CTG at onset of labour.
* Confirmation of ROM by Direct visualization or Fern test.

Exclusion Criteria:

* Contracted pelvis.
* Previous uterine surgery " upper segment ".
* Pregnancy complications like antepartum haemorrhage, pregnancy induced hypertension, gestational diabetes mellitus, IUGR.
* Fetal congenital anomalies.
* Abnormal or non reassuring fetal CTG at term or at onset of labour.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: primigravidas, full term in early labor, Ain shams maternity hospital.
Sampling Method: Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2021-10-03 (Actual); Study Completion 2021-11-20 (Actual)

PRIMARY OUTCOMES:
Incidence of cesarean section in primigravidas with unengaged fetal head in compare to primigavidas with engaged fetal head . | 24 hours
  section in primigravidas with unengaged fetal head in compare to primigavidas with engaged fetal head .

SECONDARY OUTCOMES:
Duration of labor progress in patients with unengaged | 24 Hours
  Duration of labor progress in patients with unengaged fetal head in relation to patients with engaged fetal head

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M sami, Consultant, Study Director — As.Professor
Locations (1):
- Ain Shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No